CLINICAL TRIAL: NCT04154384
Title: Life Care Specialists (LCS) With a Focus on Patient Pain Management and Prevention of Substance Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Christopher Wolf Crusade (CWC) (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mara Schenker, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00115061; CDC-IRB00115061 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2019-11-02; First posted 2019-11-06 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use
Keywords: Orthopedic surgery; Opioid addiction; Rehabilitation; Behavioral research
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methods; Referral and Consultation

STUDY DESIGN:
Intervention Model Description: There were 121 participants in the single-arm pilot trial of this study where the intervention was refined. The clinical trial portion of this study randomizes participants to receive the intervention or the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Life Care Specialist (LCS) Intervention (Experimental): In addition to receiving current standard-of-care for pain management in the aftermath of trauma, participants will have the full communication of opioid risk - via the validated Opioid Risk Tool (ORT) and a detailed substance abuse and mental health screening. As part of the daily LCS intervention, the inpatients will engage in behavioral pain management, opioid education and harm-reduction strategies (naloxone education), while also being screened for eligibility for respective referrals for complex needs, such as mental health and substance use disorders. Upon discharge, each participant will be educated by the LCS on future available modes of contact (telephone, email, video-call, follow up- visits at 2-, 6- and 12-weeks).
  Interventions: Behavioral: Life Care Specialist (LCS) Intervention
- Standard of Care with Clinical Coordination (Active Comparator): Participants will receive the current standard-of-care for pain management in the aftermath of trauma, including a standardized prescription protocol, and hospital-system approved discharge instructions which provide written instruction on how to taper opioid use and links to written/online resources for opioid misuse, overdose prevention, and State-approved disposal options.
  Interventions: Other: Clinical Coordination with Referrals
- Pilot Study of Pain Management Strategies (Other): Orthopedic trauma patients will work with a Life Care Specialist (LCS) and will receive personalized pain management strategies to avoid potential opioid misuse. Participants will be followed for one-year post-operation. An official pain management protocol will be developed during the pilot portion of this study
  Interventions: Behavioral: Pilot Study of Pain Management Strategies

INTERVENTIONS:
Behavioral: Life Care Specialist (LCS) Intervention — The Life Care Specialist (LCS) uses a two-arm approach to education by initially assessing participants general understanding of opioids upon which targeted education is tailored and applied and secondly, building a longitudinal relationship with each patient to increase the saliency of administered opioid education during postoperative follow-up. Information includes proper disposal, common symptoms of opioid use, signs of dependence and overdose and use of naloxone. Information is disseminated orally with adjunct physical resource guides including visual representations and literature.
  Other Names: Opioid Education
  Arms: Life Care Specialist (LCS) Intervention
Other: Clinical Coordination with Referrals — The Life Care Specialist (LCS) can help arrange a referral for the participant, should a medical or social issue be identified during LCS intervention, including mental health services, addiction medicine services, housing insecurity referrals, food insecurity referrals, and amputee support. When giving referrals, the LCS works closely with physicians and nurses to make sure that the participant is a good fit for the referral program.
  Arms: Standard of Care with Clinical Coordination
Behavioral: Pilot Study of Pain Management Strategies — Orthopedic trauma patients will work with a Life Care Specialist (LCS) and will receive personalized pain management strategies to avoid potential opioid misuse.
  Arms: Pilot Study of Pain Management Strategies

SUMMARY:
The overall hypothesis of this randomized-controlled trial is that the introduction of a Life Care Specialist (LCS) as a novel member of the clinical care team will help reduce opioid utilization, decrease pain scores, and improve patient understanding of their addiction risk in the aftermath of orthopaedic trauma.

DETAILED DESCRIPTION:
Opioids are psychoactive substances (narcotics) primarily used for pain relief by producing morphine-like effects. Although regularly prescribed by physicians, opioids (including morphine, codeine, and oxycodone) are highly addictive. Opioids block feelings of pain and trigger a release of dopamine. Dependence occurs with repeated use, as the parts of the brain naturally responsible for releasing dopamine rely on the drug for proper function. When avoided, patients quickly experience severe withdrawal symptoms similar to the flu.

In the United States, millions are prescribed opioids for pain relief. Every day, more than 115 people die from overdose. The highest among them are people aged 25 to 54 years. Addiction treatment costs near $78.5 billion and rising, less than 10% of people in need are receiving it.

Within the orthopaedic trauma population at Grady Healthcare in Atlanta, Georgia, 20% of patients report a history of substance abuse, 30% have previously used opioid medications for pain, and nearly 25% report taking opioid pain medications up to 1 year after their trauma. Trauma patients are particularly at high risk.

The Christopher Wolf Crusade (CWC) is a 501C3 non-profit providing preventative solutions, education, and advocacy for the American opioid epidemic. CWC's primary focus is to introduce a behavior-specific intervention at the time of inpatient hospitalization for trauma to decrease overall opioid utilization and improve pain control in the post-trauma time period. The goal of this study is to introduce the LCS to the healthcare field to focus on pain management and addiction prevention for patients. The LCS is a behavior-based pain "coach" who educates patients on risks of opioid dependence and offers non-traditional non-pharmacologic options for pain control. In addition, the LCS will act as a liaison between the patient and the physician to ensure that traditional pharmacologic-based pain control regimens are optimized.

The pain management protocol was refined through a pilot, single-center study where the LCS provided personalized pain management strategies to patients combating pain. Participants in the single-arm pilot portion of the study were enrolled beginning in February 2020 and data collection for these 121 participants was completed April 15, 2021.

The clinical trial portion of this study will include 200 patients who will be consented, enrolled, and randomized in a 1:1 fashion to A) receive the current standard-of-care for pain management in the aftermath of trauma or B) additional LCS intervention. All participants will have the same quantity and quality of interaction with their usual clinical providers and will be followed in the orthopaedic trauma clinic at routine post-operative intervals (2 weeks, 6 weeks and 3 months post-operatively).

ELIGIBILITY:
Inclusion Criteria for Single-Arm Pilot Portion of this Study:

* Orthopaedic trauma patients with planned surgical procedure
* Informed consent obtained

Exclusion Criteria for Single-Arm Pilot Portion of this Study:

* Enrolled in a study that does not permit co-enrollment
* Unlikely to comply with the follow-up schedule
* Unable to converse, read or write English or Spanish at elementary school level

Inclusion Criteria for Clinical Trial Portion of this Study:

* Orthopaedic trauma patients with an isolated injury requiring surgery
* Informed consent obtained
* Functioning cellphone

Exclusion Criteria for Clinical Trial Portion of this Study:

* Enrolled in a study that does not permit co-enrollment
* Unlikely to comply with the follow-up schedule
* Unable to converse, read or write English or Spanish at elementary school level
* Unlikely to complete surveys at home, access to phone
* Unlikely to respond to opioid utilization text messaging (SMS)
* Incarcerated
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Schenker, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, individual participant data will be made available for sharing upon request from other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will be available for sharing following publication of the findings from this study until 5 years after publication.
Access Criteria: Researchers interested in accessing data should provide a description of the proposed project to Dr. Schenker at mara.schenker@emory.edu.

REFERENCES:
- [Background] Giordano NA, Seilern Und Aspang J, Baker J, Rice CW, Barrell B, Kirk L, Ortega E, Wallace M, Steck A, Schenker ML. The effect of a Life Care Specialist on pain management and opioid-related outcomes among patients with orthopedic trauma: study protocol for a randomized controlled trial. Trials. 2021 Nov 27;22(1):858. doi: 10.1186/s13063-021-05841-1. PMID 34838101
- [Result] Giordano NA, Seilern Und Aspang J, Baker J, Medline A, Rice CW, Barrell B, Kirk L, Ortega E, Wallace M, Steck A, Schenker ML. Integration of Life Care Specialists Into Orthopaedic Trauma Care to Improve Postoperative Outcomes: A Pilot Study. Pain Manag Nurs. 2022 Oct;23(5):608-615. doi: 10.1016/j.pmn.2022.03.010. Epub 2022 Apr 25. PMID 35477669
- [Result] Giordano NA, Und Aspang JS, Baker J, Holder C, Cantu N, Checo G, Rice CW, Barrell B, Wallace M, Steck AR, Schenker ML. Can Patient-centered Education and Pain Management Delivered by Coaches Improve Pain Outcomes After Orthopaedic Trauma? A Randomized Trial. Clin Orthop Relat Res. 2024 Oct 1;482(10):1858-1869. doi: 10.1097/CORR.0000000000003121. Epub 2024 May 15. PMID 38843502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Memorial Hospital in Atlanta, Georgia, USA.
Pre-assignment Details: The nature of this preliminary research began as a single-arm pilot study but due to the COVID-19 pandemic, the pilot was suspended. Instead, a two-arm Clinical Trial was commenced due to time constraints at a time when non-essential personnel, including research staff, were permitted to safely return to the fast-paced clinical environment once infection control measures were established. The outcomes of the clinical trial portion did not apply to the pilot group.
Period: Overall Study
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination | Pilot Study of Pain Management Strategies
Started | 104 | 108 | 121
Completed | 72 | 57 | 121
Not Completed | 32 | 51 | 0
Not completed — Lost to Follow-up | 24 | 33 | 0
Not completed — Withdrawal by Subject | 7 | 18 | 0
Not completed — Missing outcome data | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The nature of this preliminary research began as a single-arm pilot study but due to the COVID-19 pandemic, the pilot was suspended. Instead, a two-arm Clinical Trial was commenced due to time constraints at a time when non-essential personnel, including research staff, were permitted to safely return to the fast-paced clinical environment once infection control measures were established. The outcomes of the clinical trial portion did not apply to the pilot group.
Groups:
- Pilot Study of Pain Management Strategies: Orthopedic trauma patients will work with a LifeCare Specialist (LCS) and will receive personalized pain management strategies to avoid potential opioid misuse. Participants will be followed for one-year post-operation. An official pain management protocol will be developed during the pilot portion of this study.
- Total: Total of all reporting groups
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination | Pilot Study of Pain Management Strategies | Total
Number analyzed (Participants) | 72 | 57 | 121 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.15 (18.17) | 42.46 (16.97) | 38.82 (15.00) | 42.84 (17.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 33 | 52 | 124
  Male | 33 | 24 | 69 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 53 | 41 | 94 | 188
  White | 17 | 15 | 12 | 44
  More than one race | 0 | 0 | 13 | 13
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 72 | 57 | 121 | 129

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale Average Pain Score
Description: For participants in the single-arm pilot study and in the dual-arm, clinical-trial portion of the study, daily pain within the last 24 hours was assessed using a 10-point Likert scale where 1 = no pain and 10 = severe pain. After Week 2, pain was assessed only during the follow-up visits.
Time Frame: Day 1 (during inpatient hospitalization), Week 2, Week 6, Month 3
Population: Outcomes for the pilot study participants were only collected up to Week 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pilot Study of Pain Management Strategies: Orthopedic trauma patients will work with a Life Care Specialist (LCS) and will receive personalized pain management strategies to avoid potential opioid misuse. Participants will be followed for one year post-operation. An official pain management protocol will be developed during the pilot portion of this study.
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination | Pilot Study of Pain Management Strategies
Number analyzed (Participants) | 72 | 57 | 121
units on a scale
  Day 1 (during inpatient hospitalization) | 7.62 (2.72) | 7.94 (2.42) | 8.43 (2.80)
  Week 2: number analyzed (Participants) | 72 | 57 | 80
  Week 2 | 5.88 (2.76) | 5.64 (2.93) | 4.74 (2.68)
  Week 6: number analyzed (Participants) | 72 | 57 | 0
  Week 6 | 4.36 (2.91) | 4.14 (3.27) |
  Month 3: number analyzed (Participants) | 72 | 57 | 0
  Month 3 | 3.79 (3.09) | 3.72 (3.16) |

2. Primary Outcome: Number of Participants With Improvement in the Numeric Rating Scale (NRS) Average Pain Score
Description: The number of participants in the dual-arm, clinical-trial portion of the study reporting a decrease in the NRS average pain score at 3 months follow-up compared to the baseline visit.
Time Frame: Month 3
Population: This outcome applies to the clinical trial groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
Participants | 64 | 42
Statistical Analysis 1: Comparison: Life Care Specialist (LCS) Intervention vs Standard of Care With Clinical Coordination; Test type: Superiority — A comparison of the proportion of participants in each arm reporting an improvement in average pain score on the Numeric Rating Scale from baseline to 3 months follow-up; p = 0.035, Chi-squared — A comparison of the proportion of participants in each arm reporting an improvement in average pain score on the Numeric Rating Scale from baseline to 12 weeks follow-up

3. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form Score
Description: For participants in the dual-arm, clinical trial portion of the study, severity of insomnia, sleep disruption, and sleep quality over the past seven days is assessed with the 4-item PROMIS Sleep Disturbance - Short Form. Responses are given on a 5-point Likert scale where 1 is equivalent to best possible and 5 is equivalent to worst possible. Raw scores are converted to t-scores ranging from 0 to 100, with a mean of 50 and standard deviation of 10. Scores below 50 indicate better sleep than the average person.
Time Frame: Day 1 (during inpatient hospitalization), Week 2, Week 6, Month 3
Population: This outcome applies to the clinical trial groups.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
T-score
  Day 1 (during inpatient hospitalization) | 52.89 (10.70) | 51.57 (10.21)
  Week 2 | 60.16 (8.69) | 58.85 (9.56)
  Week 6 | 54.74 (11.26) | 53.81 (11.56)
  Month 3 | 52.68 (11.92) | 51.28 (13.13)

4. Primary Outcome: PROMIS Pain Interference - Short Form Score
Description: For participants in the dual-arm, clinical trial portion of the study, self-reported pain interference with activities is assessed with the PROMIS Pain Interference - Short Form. Responses to the 4 items are given on a 5-point Likert scale from 1 (no interference) to 5 (much interference). Raw scores are converted to t-scores ranging from 0 to 100, with a mean of 50 and standard deviation of 10. Scores above 50 indicate worse pain interference than the average person.
Time Frame: Day 1 (during inpatient hospitalization), Week 2, Week 6, Month 3
Population: This outcome applies to the clinical trial groups only.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
T-score
  Day 1 (during inpatient hospitalization) | 54.14 (12.17) | 56.24 (11.52)
  Week 2 | 65.19 (6.37) | 65.99 (7.16)
  Week 6 | 62.28 (8.59) | 59.36 (7.93)
  Month 3 | 58.89 (10.54) | 58.19 (9.27)

5. Primary Outcome: PROMIS Physical Function - Short Form Score
Description: For participants in the dual-arm, clinical trial portion of the study, self-reported capability to conduct physical activity is assessed with the PROMIS Physical Function - Short Form. Responses to the 4 items are given on a 5-point Likert scale where 1 = unable to do and 5 = without any difficulty. Raw scores are converted to t-scores ranging from 0 to 100, with a mean of 50 and a standard deviation of 10. Scores above 50 indicate better physical function than the average person.
Time Frame: Day 1 (during inpatient hospitalization), Week 2, Week 6, Month 3
Population: This outcome applies to the clinical trial groups only.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
T-score
  Day 1 (during inpatient hospitalization) | 42.85 (13.75) | 42.31 (13.14)
  Week 2 | 26.56 (5.27) | 26.82 (6.55)
  Week 6 | 30.33 (7.31) | 33.59 (8.43)
  Month 3 | 37.22 (8.43) | 37.53 (8.00)

6. Secondary Outcome: Opioid Utilization
Description: For participants in the single-arm pilot study, and in the dual-arm, clinical-trial portion of the study, opioid utilization during inpatient hospitalization was recorded in daily morphine milligram equivalents.
Time Frame: Day 1 (during inpatient hospitalization)
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination | Pilot Study of Pain Management Strategies
Number analyzed (Participants) | 72 | 57 | 121
milligrams | 22.52 [22.50 to 30.00] | 30.00 [22.50 to 30.00] | 39.77 [25.00 to 49.82]

7. Secondary Outcome: Opioid Literacy Tool (OLT) Score
Description: For participants in the dual-arm, clinical trial portion of the study, accuracy of knowledge about opioids (3 questions) and opioid-related risks (5 questions) is assessed with an Opioid Literacy Tool (OLT). Accuracy of opioid knowledge responses are given on a dichotomous scale (yes/no). Responses for accuracy of knowledge about opioid-related risks are given on a 7-point scale where 1 = definitely true and 7 = definitely false. The score is reported as the percent of correct responses.
Time Frame: Day 1 (during inpatient hospitalization), Month 3
Population: This outcome applies to the clinical trial groups only.
Measure: Mean (Standard Deviation); unit: percentage out of 100%
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
percentage out of 100%
  Day 1 (during inpatient hospitalization) | 32.02 (27.50) | 32.69 (31.37)
  Month 3 | 33.20 (34.63) | 31.25 (33.32)

8. Secondary Outcome: Total Sleep Time
Description: For participants in the dual-arm, clinical trial portion of the study, wrist-actigraphy devices captured continuous postoperative functional outcomes among patients during their hospitalization and up to 72 hours postoperatively. Total sleep time is assessed in minutes of sleep per night.
Time Frame: Up to 72 hours (during inpatient hospitalization)
Population: This outcome applies to the clinical trial groups only. Only participants who wore the sleeping tracking device were included in this outcome.
Measure: Mean (Standard Deviation); unit: minutes/night
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 63 | 56
minutes/night | 267.34 (99.71) | 236.95 (55.6)

9. Secondary Outcome: Percentage of Sleep Fragmentation
Description: For participants in the dual-arm, clinical trial portion of the study, wrist-actigraphy devices captured continuous postoperative functional outcomes among patients during their hospitalization. The percentage of sleep fragmentation is assessed as the number of awakenings and sleep stage shifts divided by the total sleep time *100.
Time Frame: Day 1 (during inpatient hospitalization)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of sleep fragmentation
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 63 | 56
percentage of sleep fragmentation | 33.77 (15.29) | 32.68 (15.17)

10. Secondary Outcome: Patient Satisfaction Survey
Description: For participants in the dual-arm, clinical-trial portion of the study, patient satisfaction with clinical care was assessed with a modified Press Ganey Integrated Survey. This survey captured a comprehensive picture of each participant's care experience. Participants were asked "Using any number from 0 to 10, where 0 is the worst hospital possible and 10 is the best hospital possible, what number would you use to rate this hospital during your stay?" Higher scores indicate higher satisfaction.
Time Frame: Week 2
Population: This outcome applies to the clinical trial groups only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
units on a scale | 7.77 (2.39) | 7.23 (2.36)

11. Secondary Outcome: Number of Pilot Study Participants Reporting Satisfaction With Clinical Care
Description: For participants in the single-arm pilot study, patient satisfaction with clinical care was assessed by asking: "Did you find the interactions with the Life Care Specialist, (LCS) helpful in managing your pain?" Response choices ranged from "strongly agree" to "strongly disagree". Responses were dichotomized as finding the LCS helpful or not finding the LCS helpful with managing pain.
Time Frame: Week 2
Population: This analysis includes participants in the pilot group who attended their 2 weeks post-operative follow-up appointment.
Measure: Count of Participants; unit: Participants
Groups:
- Pilot Study of Pain Management Strategies Intervention: Orthopedic trauma patients will work with a Life Care Specialist (LCS) and will receive personalized pain management strategies to avoid potential opioid misuse. Participants will be followed for one-year post-operation. An official pain management protocol will be developed during the pilot portion of this study.
Arm/Group | Pilot Study of Pain Management Strategies Intervention
Number analyzed (Participants) | 80
Participants | 79

12. Secondary Outcome: Patient Assessment of Constipation-Symptoms (PAC-SYM) Score
Description: For participants in the dual-arm, clinical-trial portion of the study, the PAC-SYM instrument was used to assess the severity of patient-reported symptoms of constipation. The instrument includes 12 items with subscales assessing abdominal, rectal, and stool symptoms. Responses are given on a 5-point scale ranging from 0 (symptom absent) to 4 (very severe symptoms). The total score is calculated as the mean of all response and ranges from 0 to 4, where lower scores indicate lower symptom burden.
Time Frame: Week 2
Population: This outcome applies to the clinical trial groups only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
score on a scale | 0.49 (0.74) | 0.79 (0.76)

13. Secondary Outcome: Defense and Veterans Pain Rating Scale Score
Description: The Defense and Veterans Pain Rating Scale is a patient-reported outcome used to measure the degree to which pain influenced a respondent's ability to function over the prior 24 hours. Scores range from 0 to 10 with higher scores indicating impaired functioning due to pain.
Time Frame: Day 1 (during inpatient hospitalization), Week 2, Week 6, Month 3
Population: This outcome applies to the clinical trial groups only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination
Number analyzed (Participants) | 72 | 57
score on a scale
  Day 1 (during inpatient hospitalization) | 6.84 (3.04) | 7.49 (2.67)
  Week 2 | 5.35 (2.82) | 5.54 (2.69)
  Week 6 | 4.13 (2.76) | 4.02 (3.09)
  Month 3 | 3.68 (2.95) | 3.56 (3.25)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time consent to participate in the study was given through 90 days post-surgery.
Arm/Group | Life Care Specialist (LCS) Intervention | Standard of Care With Clinical Coordination | Pilot Study of Pain Management Strategies
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/57 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/57 | 0/121
Other Adverse Events (participants affected / at risk) | 0/72 | 0/57 | 0/121

LIMITATIONS AND CAVEATS:
The nature of this preliminary research began as a single-arm pilot study but due to the coronavirus disease 2019 (COVID-19) pandemic, the pilot was suspended. A two-arm clinical trial was commenced due to time constraints at a time when non-essential personnel, including research staff, were permitted to safely return to the fast-paced clinical environment once infection control measures were established. Many of the outcome measures for the clinical trial did not apply to the pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT04154384/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT04154384/ICF_001.pdf